CLINICAL TRIAL: NCT06333600
Title: Efficacy and Safety of Topical Vitamin D Analogue in Treatment of Female Pattern Hair Loss
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doaa Gaber Abdel baset, Assistant Lecturer, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-23-07-05
Record Dates: First submitted 2024-03-04; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Dermatology; Female Pattern Baldness
MeSH Terms: conditions — Alopecia | interventions — Minoxidil; Vitamin D; calcipotriene; Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group minoxidil (Treatment group) (Active Comparator): Topical application of Minoxidil 5% solution
  Interventions: Drug: Topical minoxidil
- Group calcipotriol (Treatment group) (Active Comparator): Topical application of vitamin D3 analogue (Calcipotriol ointment)
  Interventions: Drug: Topical Vitamin D
- Group 3 (Negative control group) (Placebo Comparator): This group will be given saline
  Interventions: Drug: Saline spray

INTERVENTIONS:
Drug: Topical minoxidil — Therapeutic intervention
  Other Names: Rogaine
  Arms: Group minoxidil (Treatment group)
Drug: Topical Vitamin D — Therapeutic intervention
  Other Names: Calcipotriol
  Arms: Group calcipotriol (Treatment group)
Drug: Saline spray — placebo
  Other Names: saline
  Arms: Group 3 (Negative control group)

SUMMARY:
The trial aims to study efficay of topical vitamin D analogue in treatment of female pattern hair loss cases

DETAILED DESCRIPTION:
Study approval: The study will be approved by Research and Ethical committee at Faculty of Medicine, Sohag University. Informed written consent will be obtained from all participants after explanation of nature of the study.

Study design: A prospective, randomized, controlled clinical study. Study population: The study will include 45 females aged 15-70 years attending Dermatology outpatient clinic at Sohag University Hospital with a complaint of chronic diffuse hair loss diagnosed clinically and will be confirmed by trichoscope as FPHL and with serum vitamin D deficiency.

Exclusion criteria will include:

* Patients with other hair loss disorders as telogen effluvium, anagen effluvium, alopecia areata, cicatricial alopecia and trichotillomania.
* Oral or parentral vitamin D supplementation for the last 3 months
* Treatment with topical vitamin D analogs in the past month
* Patients who received hair tonics or any specific hair therapy over the last 3 months prior to enrollement in the study.
* Patients with diabetes mellitus, renal disease, thyroid and parathyroid abnormalities, or autoimmune diseases.
* Patients who are pregnant, lactating or on contraceptive pills.

All patients in this study will be subjected to:

1. Complete history including:

   * Personal history: age, occupation, residence, marital status, special habits of medical importance
   * Menstrual and obstetric history
   * Average time spent outdoor (per hour)
   * Diatery habits
   * Family history of similar condition
   * History of any chronic illness or hormonal abnormalities such as hirsutism, PCO…..
   * History of hair loss including: age of onset, course, duration, affected site and any previous treatment taken by the patient and its response.
2. Hair examination will include:

   * Pattern of hair loss (Ludwig, Olsen or Norwood)
   * Pull test
   * Scalp skin condition
   * Grading according to Sinclair scale
3. Evaluating tools:

   * Gross photos will be taken under adequate illumination, identical settings, lighting, and position before starting treatment and at monthly follow up visits.
   * Trichoscopic examination: All cases will be viewed trichoscopically from frontal, temporal, and occipital views (before treatment and at follow up visits) and will be evaluated by two blinded investigators. Establishing the diagnosis of FPHL will be done according to diagnostic criteria of FPHL. Hair density, hair diameter and peripilar sign will be recorded before and after treatment.
   * Subject assessment: A 7-point scale will be used Investigations:-
   * Serum vit.D will be measured for all participants • Other investigations will be done if needed according to primary patient evaluation: CBC, serum ferritin, serum calcium level, serum creatinine, hormonal (TSH, FSH, LH, prolactin, testosterone).

Therapeutic interventions:- 45 patients diagnosed as FPHL with decreased serum vitamin D will be randomly divided into 3 treatment groups:

* Group 1 (15 patients) will apply topical 5% minoxidil solution in a dose of 1ml twice daily.
* Group 2 (15 patients) will apply topical vit. D analogue (calcipotriol ointment 0.005%) twice daily (1 fingertip unit for every 2% of body surface area)
* Group 3 (15 patients) ( placebo group).
* Any side effects will be registered such as itching, scalling, burning sensation, dryness….
* Duration of treatment will continue for 3 months

ELIGIBILITY:
Inclusion Criteria:

* All females with FPHL aging 15 - 60 years

Exclusion Criteria:

* Patients with other hair loss disorders as telogen effluvium, anagen effluvium, alopecia areata, cicatricial alopecia and trichotillomania.

  * Patients with normal serum vit.D level
  * Oral or parentral vitamin D supplementation for the last 3 months
  * Treatment with topical vitamin D analogs in the past month
  * Patients who received hair tonics or any specific hair therapy over the last 3 months prior to enrollement in the study.
  * Patients with diabetes mellitus, renal disease, thyroid and parathyroid abnormalities, or autoimmune diseases.
  * Patients who are pregnant, lactating or on contraceptive pills.

Ages: 15 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-05-20 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
Change of Sinclaire grading of Female pattern hair loss | 3 months
  clinical grading of female pattern hair loss
Change of Trichoscopic parameters (Hair dermoscopy) | 3 months
  Measure specific findings of female pattern hair loss diagnosis and follow up after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Essam A Nada, MD, Study Chair — Professor
Locations (1):
- Facult of Medicine, Sohag Uniiversity, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No